CLINICAL TRIAL: NCT04199780
Title: tDCS Combined With a Brief Cognitive Intervention to Reduce Perioperative Pain and Opioid Requirements in Veterans
Brief Title: Effects of tDCS Combined With CBI on Postsurgical Pain
Acronym: tDCS-CBI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NURB-001-19S; CX001996 (Other Grant/Funding Number: Charleston CSR&D)
Record Dates: First submitted 2019-12-06; First posted 2019-12-16 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Total Knee Arthroplasty (Postoperative Pain); Total Hip Arthroplasty (Postoperative Pain)
Keywords: total knee arthroplasty; pain; postsurgical pain; opioid; transcranial direct current stimulation; tDCS; brain stimulation; total hip arthroplasty; TKA; THA
MeSH Terms: conditions — Pain, Postoperative; Pain | interventions — Transcranial Direct Current Stimulation; Methods

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Group 1- real tDCS and real CBI (Experimental): 4 active treatments of tDCS and active cognitive behavioral intervention (CBI)
  Interventions: Device: Transcranial Direct Current Stimulation; Behavioral: Cognitive-Behavioral (CB) intervention
- Group 2- real tDCS and sham CBI (Experimental): 4 active treatments of tDCS and education-only-control cognitive intervention
  Interventions: Device: Transcranial Direct Current Stimulation; Behavioral: Cognitive-Behavioral (CB) intervention
- Group 3- sham tDCS and real CBI (Experimental): 4 sham treatments of tDCS and active cognitive behavioral intervention (CBI)
  Interventions: Device: Transcranial Direct Current Stimulation; Behavioral: Cognitive-Behavioral (CB) intervention
- Group 4- sham tDCS and sham CBI (Sham Comparator): 4 sham treatments of tDCS and education-only-control cognitive intervention
  Interventions: Device: Transcranial Direct Current Stimulation; Behavioral: Cognitive-Behavioral (CB) intervention

INTERVENTIONS:
Device: Transcranial Direct Current Stimulation — Transcranial direct current stimulation (tDCS), stimulates specific areas of the brain via electric current passed through electrodes placed on the scalp. During tDCS, low amplitude direct currents penetrates the skull to enter the brain and modulates neuronal activity.
  Other Names: tDCS
Behavioral: Cognitive-Behavioral (CB) intervention — CBI generally consist of cognitive coping strategies (e.g., distraction, relabeling, reducing pain-catastrophizing) and self-management (e.g., relaxation strategies, guided imagery) designed to enhance perceived control and reduce sympathetic nervous system tone.
  Other Names: CBI

SUMMARY:
The purpose of this study is to determine whether a new medical technology can help reduce post-operative total knee or hip pain when combined with a Cognitive-Behavioral intervention (CBI).

This new medical technology, is called transcranial direct current stimulation (tDCS), it uses a very small amount of electricity to temporarily stimulate specific areas of the brain thought to be involved in pain reduction. The electrical current passes through the skin, scalp, hair, and skull and requires no additional medication, sedation, or needles.

This study will investigate the effects of tDCS, the Cognitive-Behavioral (CB) intervention and their combination on pain among veterans following total knee arthroplasty (TKA) or total hip arthroplasty (THA). The Veteran may benefit in the form of decreased pain and opioid requirements following knee or hip replacement surgery. However, benefit is only likely if Veterans are randomized to one of the 3 (out of 4) groups.

This study hopes to determine the effects of these interventions and combined effect on post-operative pain, opioid use and functioning during the 48-hour post-operative period following a total knee or hip replacement.

DETAILED DESCRIPTION:
The proposed study employs a randomized, double-blind, sham-controlled design to evaluate the effects of tDCS, brief Cognitive-Behavioral (CB) intervention and their combination on pain among veterans undergoing unilateral TKA or THA. 132 patients undergoing TKA/THA will be randomly assigned to one of four groups:

1. Group1- real tDCS + real CB intervention
2. Group2- real tDCS + education-only-control intervention
3. Group3- sham tDCS + real CB intervention
4. Group4- sham tDCS +education-only-control intervention

Participants will receive 2 tDCS/CBI treatments on the day of their surgery, and 2 tDCS/CBI treatments the day after their surgery. Participants' perioperative medication usage and pain ratings will be tracked during postoperative hospital stay. Follow-up data regarding pain and opioid use will be collected at 1, 3 and 6-months.

ELIGIBILITY:
Inclusion Criteria:

Participants will be 120 patients (132 recruited to account for 10% drop-out rate) undergoing TKA or THA surgery at the Ralph H. Johnson VAMC in Charleston SC.

* Mentally capable of reading, writing, giving consent, and following instructions
* Cleared for, and scheduled for unilateral TKA or THA surgery
* Able to hear CB intervention and understand educational materials through headphones in English

Exclusion Criteria:

* implanted medical devices above the waist
* pregnant
* history of seizures
* allergic to latex rubber
* psychiatric conditions except for depression and/or anxiety disorders (commonly seen in this population).

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2021-01-11 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
postoperative opioid pain medication use | 48 hours
  Patient controlled analgesic medication usage (the morphine equivalent dose (MED); mg of morphine) during the acute 48-hour post-operative period following total knee arthroplasty (TKA) or total hip arthroplasty (THA).

SECONDARY OUTCOMES:
Long term outcomes of patient reported pain ratings | 1 month
  long-term outcomes of post-operative tDCS and a cognitive-behavioral intervention on pain rating assessed using a visual analog scale.
Long term outcomes of patient reported pain ratings | 3 months
  long-term outcomes of post-operative tDCS and a cognitive-behavioral intervention on pain rating assessed using a visual analog scale (minimum value =0, no pain at all; maximum value =10, worst pain imaginable).
Long term outcomes of patient reported pain ratings | 6 months
  long-term outcomes of post-operative tDCS and a cognitive-behavioral intervention on pain rating assessed using a visual analog scale (minimum value =0, no pain at all; maximum value =10, worst pain imaginable).

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey J Borckardt, PhD, Principal Investigator — Ralph H. Johnson VA Medical Center, Charleston, SC
Locations (1):
- Ralph H. Johnson VA Medical Center, Charleston, SC, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No